CLINICAL TRIAL: NCT06115005
Title: Treatment of Challenging Macular Holes Using Plasma Rich in Growth Factors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hossam Mohamed Moharram, Professor Doctor, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 360:2022
Record Dates: First submitted 2023-08-26; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations | interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Plasma rich in growth factors ( PRGF ) — Plasma rich in growth factors (PRGF) is characterized by a moderate concentration of platelets, in the absence of leukocytes.
  This absence of leukocytes is based on the fact that they synthesize matrix metalloproteinases, free radicals, and proinflammatory cytokines, which do not contribute and even impair the altered tissue regeneration

SUMMARY:
Aim of the Study:To report the structural and visual outcomes of plasma rich in growth factors in closure of challenging macular holes

DETAILED DESCRIPTION:
Challenging full thickness macular holes ( FTMH) include :

Recurrent FTMH Persistent (refractory) FTMH Macular holes in eyes with pathological myopia Large macular holes with an inner diameter of more than 650 µm. Plasma rich in growth factors (PRGF) is characterized by a moderate concentration of platelets, in the absence of leukocytes.

This absence of leukocytes is based on the fact that they synthesize matrix metalloproteinases, free radicals, and proinflammatory cytokines, which do not contribute and even impair the altered tissue regeneration Aim of the Study:To report the structural and visual outcomes of plasma rich in growth factors in closure of challenging macular holes

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Challenging FTMH which include Recurrent macular holes Persistent(refractory) macular holes Macular holes in eyes with pathological myopia Large macular holes with an inner diameter of more than 650 µm

Exclusion Criteria:

* 1-Corneal opacities 2-Glaucomatous patients 3-Co-existing macular pathology ( e.g. diabetic retinopathy, vein occlusion and age related macular degeneration ) 4-History of PPV for any reason other than FTMH

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that revealed closure of challenging macular holes | 6 months
  By clinical examination and OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University Hospital, Minya, Egypt

REFERENCES:
- [Background] Mahmoud TH, Thompson JT. The Treatment of Difficult Macular Holes. Ophthalmol Retina. 2021 Apr;5(4):315-316. doi: 10.1016/j.oret.2021.02.002. No abstract available. PMID 33814043
- [Background] Arias JD, Hoyos AT, Alcantara B, Sanchez-Avila RM, Arango FJ, Galvis V. PLASMA RICH IN GROWTH FACTORS FOR PERSISTENT MACULAR HOLE: A PILOT STUDY. Retin Cases Brief Rep. 2022 Mar 1;16(2):155-160. doi: 10.1097/ICB.0000000000000957. PMID 31895724